CLINICAL TRIAL: NCT03586440
Title: Effect of Forward Head and Rounded Shoulder Posture on Hand Grip Strength in Asymptomatic Young Adults
Acronym: FHRSP-RS-FHP
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Mohammad Mohammad Mosaad, professor of physical therapy, Cairo University
Other Study IDs: 69660304110
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Muscle Weakness
Keywords: RS-FHRSP-grip strength
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rounded shoulder posture group: -distance between the on table and posterior aspect of lateral part of acromion process ≥ 2.5 cm
- forward head rounded shoulder posture: * craniovertebral angle (CVA) ≤ 50 degree
  * distance between on table and acromion ≥ 2.5 cm
- normal posture group: 1. Craniovertebral angle> 50 degree
  2. distance between on table and acromion < 2.5 cm

SUMMARY:
* see if there is significant difference between subjects with forward head rounded shoulder posture and subjects with normal posture in hand grip strength in asymptomatic young adults
* see if there is significant difference between subjects with rounded shoulder posture and subjects with normal posture in hand grip strength in asymptomatic young adults

DETAILED DESCRIPTION:
* in forward head posture there is flexion in lower cervical vertebrae that causes tension on lower cervical nerve roots according to Harrison systemic review and these lower cervical nerve roots supply hand muscles
* also in rounded shoulder posture there is weakness in scapular stabilizers and retractors which affect proximal stability of the arm
* proximal stability is important for distal mobility
* so from this biomechanical point of veiw we conduct this study to see if forward head and rounded shoulder posture can affect hand grip strength in asymptomatic young adults.

ELIGIBILITY:
Inclusion Criteria:

66 subjects from both genders sedentary life.

* 22 subjects with rounded shoulder posture with the distance between on the table and the posterior aspect of lateral part of acromion process ≥ 2.5 cm
* 22 subjects with forward head rounded shoulder posture with craniovertebral angle ≤ 50 and the distance between on the table and the posterior aspect of lateral part of acromion process ≥ 2.5 cm
* 22 subjects with normal posture
* asymptomatic participants
* age range from 19-24 years old
* normal body mass index
* right handed subjects

Exclusion Criteria:

* • Neck or shoulder symptoms

  * Shoulder fracture
  * Shoulder dislocation
  * radiculopathy
  * Recent shoulder surgery
  * athletes
  * musculoskeletal abnormalities

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: asymptomatic young adults students
  1. forward head rounded shoulder posture group
  2. rounded shoulder posture group
  3. normal posture group
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
hand grip strength | 6 minutes
  hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: dalia M mosaad, professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy-Cairo University, Giza, Egypt